CLINICAL TRIAL: NCT02129374
Title: Direct Repair Surgery for Spondylolysis of Lumbar in Young Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin S. Yeom, Associated Professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DR-001
Record Dates: First submitted 2014-04-30; First posted 2014-05-02 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: Spondylolysis
Keywords: Spondylolysis; Lumbar spine; Young population; Direct repair; Union rate; Functional outcome
MeSH Terms: conditions — Spondylolysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Direct repair of pars defect (Experimental): The pars defect was repaired with 4.5mm cortical screw.
  Interventions: Procedure: Direct repair of pars defect
- Conservative treatment (No Intervention): The pars defect of spondylolysis was not repaired with cortical screw.

INTERVENTIONS:
Procedure: Direct repair of pars defect — Direct repair at pars defect was performed with 4.5mm cortical screw in young spondylolytic patients.
  Other Names: 4.5mm cortical screw
  Arms: Direct repair of pars defect

SUMMARY:
Lumbar spondylolysis is a relatively common condition that causes severe and perennial back pain in young populations. Conservative treatment of this condition may be futile, and may eventually require surgical treatment such as direct repair of pars defect and a segmental lumbar fusion with an anterior or posterior approach. Recently, of surgical treatment methods for spondylolysis, direct repair surgery of pars defect has been focused due to its inherited strengths. Most importantly, fusion surgery caused the affected segment to lose the nature range of motion and furthermore adjacent segment to be adversely affecting such as adjacent disc disease or degeneration, while direct repair theoretically could preserve the motion of the affected segment, which do not cause the adjacent segment problems as being the fusion surgery, as well as could produce better surgical outcomes with relatively less invasive technique as compared to fusion surgery. Moreover, previous articles have demonstrated that the direct repair surgery for spondylolysis of lumbar spine could achieve great functional and radiological outcomes. However, most of the previous studies was conducted using lower level designed study such as retrospective and small sample size, thereby prior literature does not provide clear information on the therapeutic outcome of direct repair for lumbar spondylolysis, especially for managing spondylolysis of young population.

Therefore, The investigators aimed to evaluate and determine the outcomes of direct repair surgery for lumbar spondylolysis in young population. To our knowledge, this is the first report that describes the functional and radiological outcomes of direct repair for spondylolysis in young populations with prospective cohort study design and relatively large sample size.

ELIGIBILITY:
Inclusion Criteria:

* patients for whom conservative treatment for six months and three-times injection treatments had failed
* a follow-up period of one year or more after surgery

Exclusion Criteria:

* patients with abnormal muscle activity or ambulation such as parkinsonism and neuromuscular disease.
* patient inability to accurately record results of preoperative and postoperative questionnaires due to problems such as a history of stroke, dementia, or major medical illness that required intensive treatment
* patient follow-up was limited to one year or less

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 163 (Actual)
Dates: Start 2014-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Union rate using dynamic radiographs and CT scans | Postoperative 1 year
  union rate at postoperative 1 year was evaluated using dynamic radiographs and computed tomography (CT) scans.

SECONDARY OUTCOMES:
Pain intensity on VAS | postoperative 3 months
  Pain intensity on lower back was evaluated with 10-point visual analogue scale (VAS) at the postoperative 6 months.
Pain intensity on VAS | postoperative 6 months
  Pain intensity on lower back was evaluated with 10-point visual analogue scale (VAS) at the postoperative 6 months.
Pain intensity on VAS | postoperative 12 months
  Pain intensity on lower back was evaluated with 10-point visual analogue scale (VAS) at the postoperative 6 months.
Functional outcome on ODI and SF-12 | Postoperative 3 months
  Functional outcome using oswestry disability index (ODI) and 12-item short form health survey (SF-12) was evaluated separately at the postoperative 3 months.
Functional outcome on ODI and SF-12 | Postoperative 6 months
  Functional outcome using oswestry disability index (ODI) and 12-item short form health survey (SF-12) was evaluated separately at the postoperative 3 months.
Functional outcome on ODI and SF-12 | Postoperative 12 months
  Functional outcome using oswestry disability index (ODI) and 12-item short form health survey (SF-12) was evaluated separately at the postoperative 3 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Armed Forces Yangju Hospital, Yangju, Gyounggido, South Korea